CLINICAL TRIAL: NCT01247545
Title: Effect of Remote Ischaemic Preconditioning on Clinical Outcomes in Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Remote Ischaemic Preconditioning on Clinical Outcomes in CABG Surgery
Acronym: ERICCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/0303
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Heart Disease
Keywords: Remote ischemic preconditioning; Coronary artery bypass graft surgery; Cardioprotection; Clinical Outcomes
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control treatment (sham RIC) will consist of four 5-minute simulated inflations of a blood pressure cuff placed on the upper arm. The inflations will be separated by 5-minute periods when the blood pressure cuff will be deflated.
  Interventions: Procedure: Control
- Remote ischaemic conditioning (Active Comparator): Blood pressure cuff placed on upper arm and inflated to 200mmHg for 5 minutes then deflated for 5 minutes - this cycle is repeated a total of 4 times.
  Interventions: Procedure: Remote ischaemic preconditioning

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning — Blood pressure cuff placed on upper arm and inflated to 200mmHg for 5 minutes then deflated for 5 minutes - this cycle is repeated a total of 4 times.
  Arms: Remote ischaemic conditioning
Procedure: Control — Control treatment (sham RIC) will consist of four 5-minute simulated inflations of a blood pressure cuff placed on the upper arm. The inflations will be separated by 5-minute periods when the blood pressure cuff will be deflated.
  Arms: Control

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death in the UK, accounting for 124,000 deaths (2006) and costing the UK economy over £7.9 billion a year. Patients with severe CHD are usually treated by coronary artery bypass graft (CABG) surgery, the risks of which are increasing due to older and sicker patients being operated on. New treatment strategies are therefore required to improve health outcomes in these high-risk patients undergoing CABG with or without valve (CABG±valve) surgery.

The hypothesis tested in this research proposal is that remote ischaemic preconditioning (RIC), a virtually cost-free, non-pharmacological and simple non-invasive strategy for reducing the damage to the heart muscle at the time of surgery, improves health outcomes in high-risk patients undergoing CABG±valve surgery.

In this research project, 1610 high-risk patients undergoing CABG±valve surgery will be recruited via 28 UK hospitals performing heart surgery. Patients will be randomly allocated to receive either RIC or control. For RIC, a blood pressure cuff will be placed on the upper arm to temporarily deprive it of oxygen and nutrients, an intervention which has been shown in the investigators pilot studies to reduce damage to the heart muscle by up to 40% during CABG±valve surgery. The investigators will determine whether RIC can improve health outcomes in terms of better patient survival, less heart attacks and strokes, shorter hospital stay; less damage to the heart, kidney and brain during surgery; better heart function post-surgery and less chance of developing heart failure; better exercise tolerance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing CABG with or without valve surgery using blood cardioplegia
2. Patients aged 18 years and above
3. Patients with an additive Euroscore greater than or equal to 5

Exclusion Criteria:

1. Cardiogenic shock
2. Cardiac arrest on current admission
3. Pregnancy
4. Significant peripheral arterial disease affecting the upper limbs
5. Patients with significant hepatic dysfunction (Prothrombin>2.0 ratio)
6. Patients with significant pulmonary disease (FEV1<40% predicted)
7. Patients with known renal failure with a GFR<30 mL/min/1.73 m2
8. Patients on glibenclamide or nicorandil, as these medications may interfere with RIC
9. Patients recruited into another study which may impact on the ERICCA study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1612 (Actual)
Dates: Start 2010-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events | One year post-surgery
  Combined endpoint of Cardiovascular death, MI, Revascularisation and Stroke.

SECONDARY OUTCOMES:
Peri-operative myocardial injury | 72 hours peri-operative period
  72 hours area under curve serum troponin-T
LV ejection fraction | At one year
  Echo determined LV ejection fraction
Acute kidney injury | Peri-operative
  Acute kidney injury score and 24 hour area under curve serum NGAL
30 day MACCE | 30 days post surgery
  Major adverse cardiac and cerebral events 30 days post surgery
All cause death | 1 year post surgery
Length of ITU stay | ITU stay
Length of hospital stay | Until hospital discharge
Inotrope score | 72 hours post surgery
  Inotrope score after 72 hours
6 minute Walk Test | 6 weeks and 12 months post surgery
Quality of Life | 6 weeks, 3/6/9 and 12 months post surgery
  Quality of Life assessed using the EQ-5D measurement

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Hausenloy, MD PhD, Principal Investigator — University College, London
Locations (28):
- United Kingdom (28):
  - Essex Cardiothoracic Centre, Basildon, Essex
  - Royal Sussex County Hospital, Brighton, Sussex
  - Blackpool Victoria Hospital, Blackpool
  - Papworth Hospital, Cambridge
  - Cardiff & Vale University Health Board, Cardiff
  - Edinburgh Royal Infirmary, Edinburgh
  - Golden Jubilee Hospital, Glasgow
  - Harefield Hospital, Harefield
  - Castle Hill Hospital, Hull
  - Glenfield Hospital, Leicester
  - Hammersmith Hospital, London
  - Kings College London Hospital, London
  - London Chest Hospital, London
  - Royal Brompton Hospital, London
  - St Bartholomew's Hospital, London
  - St George's Hospital, London
  - St Thomas Hospital, London
  - UCLH Heart Hospital, London
  - John Radcliffe Hospital, Manchester
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle
  - Trent Cardiac Centre, Nottingham
  - Derriford Hospital, Plymouth
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Swansea Hospital, Swansea
  - Wolverhampton Hospital, Wolverhampton

REFERENCES:
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Venugopal V, Hausenloy DJ, Ludman A, Di Salvo C, Kolvekar S, Yap J, Lawrence D, Bognolo J, Yellon DM. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing cardiac surgery with cold-blood cardioplegia: a randomised controlled trial. Heart. 2009 Oct;95(19):1567-71. doi: 10.1136/hrt.2008.155770. Epub 2009 Jun 8. PMID 19508973
- [Background] Venugopal V, Laing CM, Ludman A, Yellon DM, Hausenloy D. Effect of remote ischemic preconditioning on acute kidney injury in nondiabetic patients undergoing coronary artery bypass graft surgery: a secondary analysis of 2 small randomized trials. Am J Kidney Dis. 2010 Dec;56(6):1043-9. doi: 10.1053/j.ajkd.2010.07.014. Epub 2010 Oct 25. PMID 20974511
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Derived] Hausenloy DJ, Candilio L, Evans R, Ariti C, Jenkins DP, Kolvekar S, Knight R, Kunst G, Laing C, Nicholas J, Pepper J, Robertson S, Xenou M, Clayton T, Yellon DM; ERICCA Trial Investigators. Remote Ischemic Preconditioning and Outcomes of Cardiac Surgery. N Engl J Med. 2015 Oct 8;373(15):1408-17. doi: 10.1056/NEJMoa1413534. Epub 2015 Oct 5. PMID 26436207
- [Derived] Candilio L, Malik A, Ariti C, Barnard M, Di Salvo C, Lawrence D, Hayward M, Yap J, Roberts N, Sheikh A, Kolvekar S, Hausenloy DJ, Yellon DM. Effect of remote ischaemic preconditioning on clinical outcomes in patients undergoing cardiac bypass surgery: a randomised controlled clinical trial. Heart. 2015 Feb;101(3):185-92. doi: 10.1136/heartjnl-2014-306178. Epub 2014 Sep 24. PMID 25252696
- [Derived] Hausenloy DJ, Candilio L, Laing C, Kunst G, Pepper J, Kolvekar S, Evans R, Robertson S, Knight R, Ariti C, Clayton T, Yellon DM; ERICCA Trial Investigators. Effect of remote ischemic preconditioning on clinical outcomes in patients undergoing coronary artery bypass graft surgery (ERICCA): rationale and study design of a multi-centre randomized double-blinded controlled clinical trial. Clin Res Cardiol. 2012 May;101(5):339-48. doi: 10.1007/s00392-011-0397-x. Epub 2011 Dec 21. PMID 22186969